CLINICAL TRIAL: NCT05557890
Title: Efficacy and Experience of System Constellations in Virtual Reality (VR): A Randomized Control Feasibility Study
Brief Title: System Constellations in Virtual Reality (VR)
Acronym: SYSCO-VR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Collaborators: FH Münster University of Applied Sciences (Unknown); The Witten Institute For Family Business (Unknown)
Responsible Party: Principal Investigator, Christina Hunger-Schoppe, Chair of Clinical Psychology and Psychotherapy III, University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSCO-VR
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Psychological and Systems Functioning
Keywords: Systems Constellation; Virtual Reality (VR); Feasibility Study

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- System Constellation VR-Seminar (exp. group) (Experimental): By externalising significant elements, systemic constellations render the inner image someone has of a personally important social system in a visible and tangible way to get more clarity about psycho-social conflicts to make goal-oriented changes. In this study, the method System Constellation will be applied in a Virtual Reality (VR) setting during two to three day seminars.
  Interventions: Behavioral: System Constellation VR-Seminar
- System Constellation VR-Seminar (control group) (Experimental): By externalising significant elements, systemic constellations render the inner image someone has of a personally important social system in a visible and tangible way to get more clarity about psycho-social conflicts to make goal-oriented changes. In this study, the method System Constellation will be applied in a Virtual Reality (VR) setting during two to three day seminars. Study participants randomized to this group receive the intervention (system constellations VR-seminar) 4 months after the experimental group.
  Interventions: Behavioral: System Constellation VR-Seminar

INTERVENTIONS:
Behavioral: System Constellation VR-Seminar — individual-centered intervention in a group VR-setting, duration 2 to 3 days

SUMMARY:
The purpose of this study is to investigate the efficacy of system constellations in Virtual Reality (VR) in a monocentric, single-masked randomized controlled trial.

The method of system constellations refers to an approach which integrates ideas from organizational and family systems counseling with elements from psychodrama. The constellations are conducted in a group based VR-seminar, each VR-seminar lasting two to three days.

Based on the model of a general mental health, the effects of system constellations in VR on psychological and systems functioning are explored.

It is predicted that participation in a system constellation VR-seminar changes the level of psychological and systems functioning at 4 months.

ELIGIBILITY:
Inclusion Criteria:

* agreement to participate in a 2 to 3-day system constellations VR-seminar
* agreement to be randomized into treatment group or control group (waiting condition)
* agreement not to participate in another system constellation VR-seminar or seminar until completion of study

Exclusion Criteria:

* acute suicidal tendency
* acute psychotic episode
* acute drug or alcohol intoxication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline EB-45 Score within 4 months | Baseline, 2 weeks after treatment, 4 months after treatment
  Changes in psychological well-being will be assessed using the 'Outcome Questionnaire' in its German version (EB-45). The EB-45 is a brief 45-item self report outcome/tracking instrument designed for repeated measurement of client progress through the course of psychotherapy and following termination. The scales of the EB-45 measure symptom distress, interpersonal functioning, and social role.

SECONDARY OUTCOMES:
Experience in Social Systems Questionnaire (EXIS) | Baseline, 2 weeks after treatment, 4 months after treatment
  The subjective quality of family and organizational systems will be assessed by the EXIS (Questionnaire on experiences in systems), a self-constructed questionnaire comprising 24 items.
Questionnaire for the Evaluation of Treatment Progress (FEP-2) | Baseline, 2 weeks after treatment, 4 months after treatment
  The FEP-2, 40-item self report questionnaire, measures psychological distress according to the phase model of therapeutic change as well as the interpersonal model of psychological distress.
Bern Inventory of Psychotherapy Goals (BIT-C) | Baseline, 2 weeks after treatment, 4 months after treatment
  Goal achievement will be assessed using Goal Attainment Scaling as a method for the assimilation of achievement in a number of individually set goals into a single aggregated 'goal attainment score', providing a person-centred outcome, focused on that individual's priorities. Goal attainment scaling is operationalized by an open-ended question, in which study participants descriobe their individual goals. In a second step these goals will be coded according to the Bern inventory of psychotherapy goals (BIT-C)
Incongruence Questionnaire (K-INK) | Baseline, 2 weeks after treatment, 4 months after treatment
  Motivational incongruence is defined as the unsatisfactory realization of motivational goals and is based on the concept of General Psychotherapy by Klaus Grawe. The Incongruence Questionnaire (INK) is an instrument that assesses motivational incongruence, defined as the discrepancy between a person's motivational goals and his/her perception of reality. The short version of this questionnaire that will be used in our study (K-INK) comprises 23 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Witten/Herdecke University, Witten, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunger C, Bornhauser A, Link L, Schweitzer J, Weinhold J. Improving experience in personal social systems through family constellation seminars: results of a randomized controlled trial. Fam Process. 2014 Jun;53(2):288-306. doi: 10.1111/famp.12051. Epub 2013 Nov 19. PMID 24251855
- [Background] Hunger C, Weinhold J, Bornhauser A, Link L, Schweitzer J. Mid- and long-term effects of family constellation seminars in a general population sample: 8- and 12-month follow-up. Fam Process. 2015 Jun;54(2):344-58. doi: 10.1111/famp.12102. Epub 2014 Sep 29. PMID 25264190
- [Background] Weinhold J, Hunger C, Bornhauser A, Link L, Rochon J, Wild B, Schweitzer J. Family constellation seminars improve psychological functioning in a general population sample: results of a randomized controlled trial. J Couns Psychol. 2013 Oct;60(4):601-9. doi: 10.1037/a0033539. Epub 2013 Aug 19. PMID 23957767
- [Background] Hunger C, Bornhauser A, Link L, Geigges J, Voss A, Weinhold J, Schweitzer J. The Experience in Personal Social Systems Questionnaire (EXIS.pers): Development and Psychometric Properties. Fam Process. 2017 Mar;56(1):154-170. doi: 10.1111/famp.12205. Epub 2016 Feb 8. PMID 26858173
- [Background] Hunger, C. (2020). Family constellations as single intervention within the group setting in chronic psychosocial conflicts: short-, medium-, and long-term efficacy.Zeitschrift für Psychiatrie, Psychologie und Psychotherapie, 68(4), 263-273.
- [Derived] van Bebber T, Tappe EH, Druyen T, Kleve H, Rusen T, Hunger-Schoppe C. Efficacy and experience of system constellations in virtual reality (VR): study protocol for a randomized controlled feasibility study. Pilot Feasibility Stud. 2024 Dec 12;10(1):149. doi: 10.1186/s40814-024-01513-4. PMID 39668350